CLINICAL TRIAL: NCT00731718
Title: Control of Head Lice in Children and Adults
Brief Title: Control of Head Lice Infestations in Children and Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larada Sciences, Inc. (Industry)
Responsible Party: Dale Clayton, PhD, Larada Sciences, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS/LB-001; IRB 008018
Record Dates: First submitted 2008-04-23; First posted 2008-08-11 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2008-08

CONDITIONS: Pediculosis
Keywords: Head Lice
MeSH Terms: conditions — Lice Infestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: lousebuster — Subject serves as own control the length of treatment is approximately 30 minutes for full head treatment

SUMMARY:
The goal of this study is to see if heated air will kill head lice and their eggs. The treatment visit is approximately 1 hour long with a follow up phone call.

DETAILED DESCRIPTION:
Head lice strikes fear into the hearts of parents of school age children. Ridding a child of head lice is one of the most frustrating experiences a parent can face.

The objective of this project is to test whether louse desiccation using our prototype is an effective means of controlling head louse infestations in children.

Children age 6 and over are included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 6 years old, male or female Parent to attend treatment Able to comb the hair with no problems

Exclusion Criteria:

* Chemical shampoos used within 14 days Open sores or wounds on the scalp Recent head radiation

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of using heated air to kill head lice and their eggs | Through out

SECONDARY OUTCOMES:
Safety of device | Through out

CONTACTS AND LOCATIONS:
Overall Officials: Dale Clayton, PhD/Biology, Principal Investigator — Larada Sciences Inc., University of Utah
Locations (1):
- Larada Sciences,Inc., Salt Lake City, Utah, United States

REFERENCES:
- [Background] Goates BM, Atkin JS, Wilding KG, Birch KG, Cottam MR, Bush SE, Clayton DH. An effective nonchemical treatment for head lice: a lot of hot air. Pediatrics. 2006 Nov;118(5):1962-70. doi: 10.1542/peds.2005-1847. PMID 17079567
- [Derived] Bush SE, Rock AN, Jones SL, Malenke JR, Clayton DH. Efficacy of the LouseBuster, a new medical device for treating head lice (Anoplura:Pediculidae). J Med Entomol. 2011 Jan;48(1):67-72. doi: 10.1603/me10122. PMID 21337950
- See also: National Pediculosis Association — http://headlice.org